CLINICAL TRIAL: NCT06648681
Title: A Randomized Trial of Lemborexant for the Prevention of Delirium After Cardiac Surgery (PROTEX): A Pilot Study
Brief Title: Lemborexant to Prevent Post-operative Delirium in Cardiac Surgery Patients
Acronym: PROTEX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Eisai Inc. (Industry); Providence Health Care, British Columbia (Unknown); St. Paul's Hospital, Vancouver (Providence Health Care) (Unknown)
Responsible Party: Principal Investigator, Ron Ree, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H24-00546; NOL 290159 (Other: Health Canada); NOL 294580 (Other: Health Canada)
Record Dates: First submitted 2024-10-12; First posted 2024-10-18 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Delirium - Postoperative; Cardiac Surgery; Cardiac Surgery Subjects; Orexin Antagonist; Feasibility Studies; Sleep; In-hospital Mortality
Keywords: lemborexant; Postoperative Delirium; sleep medication; ICDSC; CAM; cardiac surgery; sleep aid; open heart surgery; delirium; sleep quality; Richards-Campbell Sleep Questionnaire
MeSH Terms: conditions — Emergence Delirium; Delirium; Sleep Initiation and Maintenance Disorders | interventions — lemborexant; Population Groups

STUDY DESIGN:
Intervention Model Description: This is a single centre, randomized, double blinded, placebo-controlled pilot trial, with 1:1 allocation of study drug to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive the study drug, Lemborexant 5mg, daily for 7 days post-operatively while in hospital.
  Interventions: Drug: Lemborexant 5 mg
- Control (Placebo Comparator): The Control arm will receive the placebo study drug daily for 7 days post-operatively while in hospital.
  Interventions: Drug: Control (placebo) group

INTERVENTIONS:
Drug: Lemborexant 5 mg — The intervention is the oral administration of a study drug containing lemborexant 5 mg daily between 2000h and 0000h for the first 7 days following extubating/initiation criteria is met or until their hospital discharge or until the first diagnosis of delirium, whichever occurs first.
  Initiation criteria:
  I. The participant has been extubated for at least 2 hours II. all other sedative medications have been discontinued for >1 hour III. the participant has a Richmond Agitation and Sedation Scale (RASS) score of >-1 or a Pasero Opioid-induced Sedation Scale (POSS) score <3.
  If satisfactory sleep is not achieved with the 5 mg dose of the study drug, as defined by a Richards Campbell Sleep Score <50 within 1 hour, another insomnia medication may be administered on participant request and clinician judgement.
  If participants develop delirium, the study drug will be discontinued.
  Arms: Intervention
Drug: Control (placebo) group — The control group will receive an oral placebo tablet daily between 2000h and 0000h for the first 7 days following when initiation criteria is met or until their hospital discharge, whichever occurs first.
  Initiation criteria:
  I. The participant has been extubated for at least 2 hours II. all other sedative medications have been discontinued for >1 hour III. the participant has a Richmond Agitation and Sedation Scale (RASS) score of >-1 or a Pasero Opioid-induced Sedation Scale (POSS) score <3.
  If satisfactory sleep is not achieved with the 5 mg dose of the study drug, as defined by a Richards Campbell Sleep Score <50 within 1 hour, another insomnia medication may be administered on participant request and clinician judgement.
  If participants develop delirium, the study drug will be discontinued.
  Arms: Control

SUMMARY:
Post-operative delirium is a common complication following cardiac surgery and is associated with increased 1 year mortality. Currently there are no drug therapies to prevent delirium. Orexin is a neuromodulator thought to play an important role in disordered sleep, one of the instigators of delirium. Lembrorexant is an orexin antagonist, originally approved for sleep, that may also reduce the incidence of delirium. The Investigators propose a pilot study to determine the feasibility of a randomized controlled trial comparing Lembrorexant to placebo in patients following cardiac surgery in reducing the incidence of delirium, and improving sleep.

DETAILED DESCRIPTION:
Purpose:

This is a pilot study to determine the feasibility of a larger randomized controlled trial comparing lemborexant to placebo in patients following cardiac surgery. The primary outcome of this feasibility study is to determine the rate of enrolment, adherence and retention of patients. Secondary outcomes will include incidence of postoperative delirium, delirium days, quality of sleep, hospital length of stay, and the safety and adverse side effect profile of Lemborexant.

Hypothesis:

1) Primary outcome: It is feasible to perform a study of lembrorexant versus placebo in patients after cardiac surgery, as defined by achieving a recruitment rate of at least 70% and adherence rate of 80% to the study protocol and drug administration schedule.

Justification:

Postoperative delirium is a frequent complication after cardiac surgery, with an incidence estimated at 20-52%. It is associated with increased 1 year mortality, longer ICU and hospital length of stay, and declines in functional and cognitive status that may persist for up to one year. Orexin, a neuromodulator regulating sleep and wakefulness, is believed to significantly influence the pathophysiology of delirium through its association with disordered sleep. Thus far, there are no promising therapies in prevention or treatment of post cardiac surgery delirium.

Lemborexant is a novel orexin antagonist that has been approved for treating insomnia, and has shown promising results in some studies in reducing incidence of delirium post-cardiac surgery. However, the generalizability of these studies is limited by small numbers of patients, an exclusively Asian population, variability in clinical settings, use of different clinical delirium assessment tools, and variability in comparator groups. In addition, the safety profile of lembrorexant has not been well established in the cardiac surgery population.

Objectives:

Primary Objective: to determine the rate of enrolment, adherence and retention of patients in a randomized controlled trial comparing Lemborexant to placebo early after cardiac surgery.

Secondary Objective: to compare the incidence of postoperative delirium, quality of sleep as measured by Richard Campbell's Sleep Questionnaire (RCSQ), delirium days, hospital length of stay between Lembrorexant and placebo. To determine the safety and adverse side effect profile of Lemborexant.

Research Design:

This will be a single centre, randomized, double blinded, placebo-controlled pilot trial, with 1:1 allocation of study drug to placebo. Local enrollment local is 60 patients (30 control, 30 experimental).

Statistical Analysis plan:

Patient characteristics will be described using means and standard deviations for continuous data and proportions (%) for categorical data. All analyses will be conducted on the intention-to-treat population. For the primary feasibility outcomes, the investigators will calculate 95% confidence intervals using the whole trial sample. For the secondary outcomes, the investigators will compare proportions with Lembrorexant vs placebo two-sample t-test for parametric data and Wilcoxon Rank Sum test for non parametric data. Analyses will be conducted using R 4.0.5.

Sample Size Calculation: To assess feasibility outcomes, the sample size was calculated to estimate an adherence rate of 80% with a 95% confidence interval of +/- 10%. From this calculation, the sample size will be set at 60 participants, or 10% of the sample size of a definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital following open cardiac surgery through midline sternotomy

Exclusion Criteria:

* ● Known severe obstructive sleep apnea diagnosed by polysomnography or STOPBANG score > 5

  * Periodic limb movement disorder or restless legs syndrome
  * Narcolepsy
  * Somnolence (Pasero Opioid Sedation Scale (POSS) >2)
  * Current alcohol or substance use disorder as defined by the DSM-V
  * Patient already taking moderate or strong CYP3A inhibitors
  * Frequent use of medications for insomnia defined as >4 days per week.
  * Liver failure (Child-Pugh score B or C)
  * Renal failure (eGFR<30 ml/min/1.73 m2)
  * Pre-existing delirium (ICDSC score >3 or CAM/CAM-ICU positive) at time of consent
  * BMI>40 kg/m2
  * Known allergy or hypersensitivity to study drug
  * Inability to communicate in English

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | Prior to Surgery, for the duration of the study recruitment period, estimated to be approximately 2 years
  Recruitment will be deemed feasible if the investigators are able to achieve a minimum recruitment rate of 2 patients per week, with 80% of eligible patients approached consenting to participate.
Data Collection Adherence | Post-operative day 0 to 7
  Data collection adherence will be defined as 80% completion of delirium screening and sleep scores

SECONDARY OUTCOMES:
Incidence of Postoperative Delirium | Post-operative day 0 at baseline (immediately before administration of the drug/placebo) and every 12 hours following drug/placebo administration until end of the 7 day follow-up
  Delirium will be assessed using the screening tools ICDSC (ICU Delirium Screening Checklist) while the patient is in the Cardiac Surgery Intensive Care Unit (CSICU) and CAM (Confusion Assessment Method) when the patient is on the hospital ward. The ICDSC is an 8-item delirium screening instrument (range: 0-8 points) that evaluates a patient's level of consciousness, inattention, disorientation, hallucinations or delusions, psychomotor activity, inappropriate speech or mood, sleep disturbance and fluctuation of symptoms. The CAM is a tool that assesses for the four features of delirium: Feature 1 is an acute change in mental status or a fluctuating mental status, Feature 2, is inattention, Feature 3, is altered level of consciousness and Feature 4, is disorganized thinking. Assessors rate each feature as present or not present based on guiding questions.
Delirium Days | Post-operative day 0 to 7
  The number of days where delirium was present in the post-operative study period. Postoperative delirium is defined by either: ICU Delirium Screening Checklist (ICDSC) score >3 in the cardiac surgical ICU (CSICU) or a positive Confusion Assessment Method (CAM) score on the postoperative surgical ward. The ICDSC is an 8-item delirium screening instrument (range: 0-8 points) that evaluates a patient's level of consciousness, inattention, disorientation, hallucinations or delusions, psychomotor activity, inappropriate speech or mood, sleep disturbance and fluctuation of symptoms. The CAM is a tool that assesses for the four features of delirium: Feature 1 is an acute change in mental status or a fluctuating mental status, Feature 2, is inattention, Feature 3, is altered level of consciousness and Feature 4, is disorganized thinking. Assessors rate each feature as present or not present based on guiding questions.
Adverse side effects | At the time of study drug initiation (T0) and daily following drug/placebo administration (T1 onwards) until end of the 7 day study follow-up.
  Adverse side effects other than delirium, including daytime somnolence. Daytime somnolence will be assessed by the Pasero Opioid-Induced Sedation Scale (POSS). For every instance of a study drug discontinuation, a form will be completed documenting the clinical reasons for discontinuation.
Sleep Quality | Preoperative baseline (time of recruitment/consent T -1), and daily following drug/placebo administration (T1 onwards) until end of the 7 day follow-up.
  Sleep quality will be assessed using the Richards-Campbell Sleep Questionnaire (RCSQ) which is a validated instrument to assess sleep quality in critically ill patients. It evaluates perceptions of sleep depth, sleep latency, number of awakenings, time spent awake, and overall sleep quality. There are 5 questions with a 100 point Visual Analogue Scale with 100 being the best outcome and 0 being the worst. For example, the participant is asked to rate their sleep depth, "My sleep last night was a:" from 0 (light sleep), to 100 (deep sleep). This questionnaire will be administered by a trained member of the research team daily for the duration of administration of the study drug. The score is reported as the mean of the 5 questions.
Incidence of Additional Sleep Medications | Post-operative day 0 to 7
  Incidence of participants requiring additional sleep medications.
Postoperative Hospital Length of Stay | Postoperative day 0 until hospital discharge, usually about 5-7 days postoperatively
  Number of days a patient is in hospital postoperatively.
In-Hospital Mortality | from postoperative day 0 to hospital discharge, usually 5-7 days postoperatively
  Incidence of mortality while in hospital for their index surgery

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No